CLINICAL TRIAL: NCT00936325
Title: Studies in the Pathogenesis of Systemic Capillary Leak Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090184; 09-I-0184
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10-28

CONDITIONS: Systemic Capillary Leak Syndrome
Keywords: SCLS; Natural History; Systemic Capillary Leak Syndrome
MeSH Terms: conditions — Capillary Leak Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers: healthy volunteers to act as controls.
- Patients with SCLS: patients who have been diagnosed, or are suspected of having systemic capillary leak syndrome.
- Relatives: relatives of patients who have systemic capillary leak syndrome.

SUMMARY:
Background:

* Systemic Capillary Leak Syndrome (SCLS) is a disorder of unknown cause characterized by episodes of life-threatening drop in blood pressure and leakage of fluids into tissues. The outcome from an episode of SCLS may be mild and resolve on its own, or may be severe and result in death. Although SCLS likely involves abnormalities in the cells lining blood vessels, the specific cause(s) of this disorder are not known.
* The treatment of choice for an acute SCLS episode is intravenous fluids and drugs such as norepinephrine (adrenaline), which are given to keep blood pressure at a level that will maintain vital organ function. This may be followed by a course of intravenous steroids and IVIG. Currently, there is no cure, but IVIG has been effective in diminishing the frequency and/or intensity of SCLS episodes when given regularly, as long-term effective preventive therapy for many patients who experience recurrent episodes of SCLS.
* This protocol is focused on understanding what causes SCLS with the hope that research findings will lead to the design of safe and more effective treatments.

Objectives:

- To investigate mechanisms that may cause Systemic Capillary Leak Syndrome.

Eligibility:

* Patients between 16 and older who have been diagnosed with SCLS. Patients who have been diagnosed with SCLS and are between the ages of 7 and 16 may participate off-site, by sending specimens to the NIH. Patients 16 and older who have been diagnosed with SCLS and cannot travel to the NIH may also participate off-site.
* Patients must have a documented history of at least one episode of SCLS with all three of the following documented on at least one occasion: low blood volume, low blood pressure without cause, and evidence of protein leakage during the episode. A letter of a referral from a treating physician is also required.

Design:

* Patients seen on site will be evaluated at the National Institutes of Health (NIH) for approximately 4 to 5 days on an inpatient basis, and will undergo the following procedures:

  * Medical history and physical examination.
  * Blood samples for evaluation and research purposes, as well as possible genetic testing.
  * Apheresis procedure, if needed, to obtain a larger volume of blood cells for research.
  * Bone marrow biopsy, if medically indicated.
  * Other medically indicated tests, such as skin tests to check for possible allergic reactions.
* Patients who have a capillary leak episode while at NIH will be treated with the standard of care for treating SCLS.
* Patients will be discharged from the protocol 1 year after the NIH visit.
* Patients participating off-site will be asked to collect and send specimens (such as blood) to the NIH for research purposes and evaluation.
* Unaffected Biological relatives of SCLS patients and Unrelated Normal Volunteers may also enroll on the study. Relatives and Normal Volunteers may be asked to provide research samples for the study, such as skin biopsy and research blood specimens.

DETAILED DESCRIPTION:
The systemic capillary leak syndrome (SCLS, Clarkson syndrome) is an exceedingly rare disorder of unknown cause characterized by chronic edema or acute transient, severe episodes of hypotension, hypovolemia, and oliguria. Severe edema results from leakage of fluid and macromolecules (200-900 kDa) into tissues. Acute SCLS episodes carry a high morbidity and mortality (25-30%). Fewer than 500 cases have been reported worldwide since 1960, although the disease may be underdiagnosed due to the nonspecific nature of the presenting signs and symptoms and the considerable overlap with other shock syndromes including sepsis, anaphylaxis, and angioedema. Approximately 85% of such individuals have a monoclonal gammopathy of unknown significance (MGUS), but the relationship of this finding to disease pathogenesis is unclear. This protocol will focus on the pathogenesis of SCLS. Subjects with documented episodes of capillary leak will be evaluated in order to correlate both clinical and laboratory features that are typical of SCLS. The goal is to identify biological factors and/or genetic and molecular events that may predispose to SCLS episodes. We plan to enroll up to 270 total subjects in this study, which includes affected subjects, family members, and healthy volunteers. We anticipate that our findings may be a first step toward the development of new targeted therapies.

ELIGIBILITY:
* PARTICIPANT INCLUSION CRITERIA:

Subjects with SCLS under 8 years of age are only eligible for components of this protocol that can occur Off Site and samples can be sent to the NIH. All SCLS subjects must be at least 8 years old to participate in any other aspects of this protocol at the NIH.

Subjects with SCLS may enter study while pregnant and remain on study after becoming pregnant. At the discretion of the investigator, some components of this protocol will not occur while subject is pregnant.

Diagnosis or suspected diagnosis of Systemic Capillary Leak Syndrome by a physician or documented history of capillary leak as characterized by one or more of the following:

1. Hypotension (systolic blood pressure typically less than 90 mm Hg or diastolic blood pressure less than 60 mm Hg) or associated symptoms of hypotension (e.g., hypotonia [collapse], lightheadedness or syncope, incontinence, increased thirst)
2. Laboratory evidence of hemoconcentration (e.g., hemoglobin levels above the normal range [typically greater than17 g/dL], elevated leukocyte counts).
3. Clinical evidence of fluid extravasation (e.g. edema) and/or laboratory evidence of protein extravasation such as serum hypoalbuminemia (less than 3.5 g/dL) either chronically or during an acute hypotensive episode.

   Letter of referral, with copies of pertinent medical history and laboratory studies, from prospective study subject s referring physician. Patients may self-refer, but a letter of referral from primary physician is still required.

   Willing to donate blood for sample storage to be used for future research.

   PARTICIPANT INCLUSION CRITERIA FOR THE SUBJECT'S RELATIVES/HEALTHY VOLUNTEERS:

   Willing to donate blood for sample storage to be used for future research.

   Relatives must be at least 3 years old.

   Healthy volunteers must be at least 18 years old.

   Relatives may be pregnant or become pregnant while participating in this protocol. At the discretion of the investigator, some components of this protocol will not occur while subject is pregnant. No skin biopsies or intradermal testing will be done on pregnant relatives. Bloodwork volumes may be decreased at the discretion of the investigator.

   Healthy volunteers may not be pregnant.

   Able to give informed consent.

   PARTICIPANT EXCLUSION CRITERIA:

   Presence of conditions which, in the judgment of the investigator or the referring physician, may put the subject at undue risk for travel (including frequent episodes of severe capillary leak, symptoms not preventable by pre-medication, acute infection, severe thrombocytopenia [minimum platelet count of 30,000/(proportionaly)L], or significant cardiovascular disease)

   Any condition that in the view of the principal investigator would make the subject unsuitable for enrollment in this study, (i.e. medically unstable, unable to provide phlebotomy samples).

   There is an identified cause for hypotensive episodes and/or tissue swelling.

   PARTICIPANT EXCLUSION CRITERIA FOR THE SUBJECT'S RELATIVES/HEALTHY VOLUNTEERS:

   Presence of conditions which in the judgment of the investigator or the referring physician may put the subject at undue risk (i.e. medically unstable, unable to provide phlebotomy samples).

   Any condition that in the view of the principal investigator would make the subject unsuitable for enrollment in this study (i.e. medically unstable, unable to provide phlebotomy samples).

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2009-08-24 (Actual)

PRIMARY OUTCOMES:
Identify potential causative factors and to explore genetic and/or cellular abnormalities that correlate with clinical features of SCLS. | Patients return to NIH as necessary
  Identify causative mechanisms of SCLS that will aid in diagnosis and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk M Druey, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We would provide raw data from IP included in any publication upon request. Since we are not an interventional clinical trial, this would pertain mainly to observational studies.@@@@@@@@@@@@In general, we include all IPD in the papers themselves.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting immediately after publication
Access Criteria: IPD will be shared with professional colleague upon reasonable request for any requested analysis through secure file transfer. NIH IRB may be asked to review requests, but no specific criteria for these reviews has been identified.

REFERENCES:
- [Background] Cicardi M, Gardinali M, Bisiani G, Rosti A, Allavena P, Agostoni A. The systemic capillary leak syndrome: appearance of interleukin-2-receptor-positive cells during attacks. Ann Intern Med. 1990 Sep 15;113(6):475-7. doi: 10.7326/0003-4819-113-6-475. No abstract available. PMID 2386338
- [Background] Atkinson JP, Waldmann TA, Stein SF, Gelfand JA, Macdonald WJ, Heck LW, Cohen EL, Kaplan AP, Frank MM. Systemic capillary leak syndrome and monoclonal IgG gammopathy; studies in a sixth patient and a review of the literature. Medicine (Baltimore). 1977 May;56(3):225-39. doi: 10.1097/00005792-197705000-00004. PMID 870792
- [Background] CLARKSON B, THOMPSON D, HORWITH M, LUCKEY EH. Cyclical edema and shock due to increased capillary permeability. Am J Med. 1960 Aug;29:193-216. doi: 10.1016/0002-9343(60)90018-8. No abstract available. PMID 13693909
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-I-0184.html

DOCUMENTS (1):
  • Informed Consent Form (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT00936325/ICF_000.pdf